CLINICAL TRIAL: NCT04716140
Title: Prospective Study: The Effect on Clinical Outcome After Treatment of MTP Cartilage Lesions
Brief Title: Prospective Study: The Effect on Clinical Outcome After Treatment of MTP Cartilage Lesions in Hallux Valgus Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tom Lootens (Other)
Responsible Party: Sponsor-Investigator, Tom Lootens, Principle Investigator, Algemeen Ziekenhuis Maria Middelares
Organization: Algemeen Ziekenhuis Maria Middelares (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMS.2020.006
Record Dates: First submitted 2020-11-09; First posted 2021-01-20 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Hallux Valgus; Cartilage Damage
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MTP1 joint with no cartillage laesion or grade I (No Intervention): Patients in whom no treatment of the cartilage lesions is performed: these patients have no cartilage lesion or a grade I cartilage lesion at the MTP I joint that has been found peroperatively. The degree of the cartilage lesions will be determined on the basis of the ICRS scale and an MS Hololens.
- MTP1 joint with cartillage laesion > grade I - non treatment (No Intervention): Patients in whom a cartilage lesion> grade 1 is found during surgery randomised in the no treatment group
- MTP1 joint with cartillage laesion > grade I - treatment (Experimental): Patients in whom a cartilage lesion> grade 1 is found during surgery randomised in the treatment group. They will be treated through debridement of the lesion and microfracture.
  Interventions: Procedure: Debridement of the MTP1 cartillage lesion and microfracture

INTERVENTIONS:
Procedure: Debridement of the MTP1 cartillage lesion and microfracture — Patients with a MTP1 cartillage lesion > grade I (based on based on the ICRS scale and an MS HoloLens measurement) randomised in the treatment group will be treated with debridement and microfracture
  Arms: MTP1 joint with cartillage laesion > grade I - treatment

SUMMARY:
The aim of this study is to investigate the point or nonsense of treating cartilage lesions at the level of the first metatarsophalane joint. To date, no clear guidelines have been found in the literature with regard to the treatment of cartilage lesions at the MTP I joint during corrective surgery for hallux valgus, nor has it been investigated whether this can have an effect on the clinical outcome.

DETAILED DESCRIPTION:
A randomized, single surgeon study in which two groups will be compared with each other:

Group 1: 50 patients in whom no treatment of the cartilage lesions is performed: these patients have no cartilage lesion or a grade I cartilage lesion at the MTP I joint that has been found to be operative. The grade of the cartilage lesions will be determined on the basis of the ICRS scale and an MS Hololens.

Group 2: 50 patients with a cartilage lesion> grade 1 found during surgery. Whether or not to treat the cartilage injury will be randomly determined. 50 envelopes will be made with 25 treat, 25 not to treat. Just before surgery, Dr. T. Lootens an envelope will be drawn which will determine the further policy of the operation:

Group 2A: 25 patients who are not treated for the cartilage injury. Group 2B: 25 patients who are treated for the cartilage injury by means of debridement of the lesion and microfracture.

The patients who will undergo surgery for hallux valgus will be seen pre-operatively at the outpatient clinic by the investigators. During this consultation, an explanation will be given about the research and the participant will have to sign an informed consent before participating in the study. Here, the participant will also receive an envelope with questionnaires (AOFAS score / SF 36 score / VAS pain and satisfaction), which they will fill out on the day of surgery.

Follow up The participants will be seen again at the orthopedics outpatient clinic for clinical follow-up and filling out questionnaires at 10 days, 5 weeks, 4 months and 1 year postoperatively. This follow up will be done by the co-investigator, who is blinded during the study.

Scientific foundation Corrective hallux valgus surgery currently exists in two ways: open and closed (percutaneous) technique. To date, there is no consensus on the treatment of visible cartilage lesions at the MTP I joint during the open technique. It is not known whether or not treating these injuries has an impact on the patient's clinical outcome. The Principle investigator already treats the serious cartilage lesions (> GR1 lesions) by means of debridement of the lesion, followed by microfracture. As there is no literature available on this topic yet, this research could certainly add value for the therapeutic approach of cartilage lesions at MTP I in the future.

Moreover, if microfracture gives a significantly better clinical outcome, this means that the closed (percutaneous) technique is contraindicated as a corrective technique in patients with hallux valgus. If this is not the case, no cartilage lesions at the level of the MTP I joint need to be taken into account during open technique.

ELIGIBILITY:
Inclusion Criteria:

* hallux valgus

Exclusion Criteria:

* younger than 30 years, older than 60 years
* extra pathologies other than hallux valgus

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in AOFAS | 10 days, 5 weeks, 4 months, 1 year
  American Orthopaedic Foot and Ankle Society (AOFAS) score - combines a clinician-reported and a patient-reported part for measuring the outcome of treatment in patients who sustained a complex hindfoot injury based on pain, function and alignment: 0 (bad outcome) to 100 (very good outcome)
Change in SF36 | 10 days, 5 weeks, 4 months, 1 year
  Short Form 36 (SF-36) Health Survey - consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change in VAS pain | 10 days, 5 weeks, 4 months, 1 year
  Visual Analogue Scale pain score - 0 (no pain) to 10 (worse pain)

SECONDARY OUTCOMES:
Change in VAS Patient satisfaction | 10 days, 5 weeks, 4 months, 1 year
  Visual Analogue Scale Patient satisfaction score - 0 (not satisfied at all) to 10 (very satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Maria Middelares, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No